CLINICAL TRIAL: NCT04349254
Title: Observational Study of Vision Improvement in Late Stage Dry AMD Patients by a Low Vision Aid Device
Brief Title: Observational Study of Vision Improvement in Late Stage Dry AMD Patients
Status: Completed | Type: Observational
Sponsor: Optimal Acuity Corporation (Industry)
Collaborators: Bochner Eye Institute (Other)
Responsible Party: Sponsor
Other Study IDs: Retro1
Record Dates: First submitted 2020-04-14; First posted 2020-04-16 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Dry Age-related Macular Degeneration
Keywords: Dry AMD

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Corneal treatment by a low vision aid device — Near infrared light is used to irradiate the cornea to change the modulus of small volumes of anterior stroma. The change of modulus produces a change of corneal stiffness and shape that modifies the distribution of light onto the retina. Light rays are redirected from dysfunctional areas of the retina that have been damaged by age-related macular degeneration (AMD) to functional areas of the retina, thereby improving patient vision.

SUMMARY:
The purpose of this study is to assess the vision improvement achieved by patients with late stage dry age-related macular degeneration who received corneal treatments by a low vision aid device.

DETAILED DESCRIPTION:
The purpose of this study is to assess the vision improvement achieved by patients with late stage dry age-related macular degeneration who received corneal treatments by a low vision aid device. Patient records for patients with at least 12 months follow-up will be analyzed to determine measures of vision improvement including best spectacle-corrected distance and near visual acuity. Analyses will include descriptive statistics and correlation between outcomes and baseline characteristics.

ELIGIBILITY:
Inclusion Criteria:

1. - Male or female
2. - Any race
3. - Patient is at least 50 years old
4. - Patient has diagnosed late stage dry age-related macular degeneration in one or both eyes.
5. - Treated eyes were pseudophakic at the time of treatment.
6. - Patient had moderate to severe baseline vision impairment with best spectacle-corrected distance visual acuity (CDVA) of 20/63 or worse (decimal = 0.317 or less; logMAR greater than or equal to 0.50) in the treated eye(s).
7. - Patient CDVA records are available at baseline and at 12 month post-treatment.

Exclusion Criteria:

1. - Corneal disease or disorder in either eye.
2. - Increased intraocular pressure (above 20 mm Hg), glaucoma or history of glaucoma.
3. - Presence or history of any other condition or finding that, in the opinion of the investigator, makes the patient unsuitable for retrospective observational study.

   -

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with vision impairment due to late stage dry age-related macular degeneration.
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2020-08-14 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
CDVA | 12 months
  Best spectacle-corrected distance visual acuity (CDVA)

SECONDARY OUTCOMES:
CNVA | 12 months
  Best spectacle-corrected near visual acuity (CNVA)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Berry, PhD, Principal Investigator — Optimal Acuity Corporation
Locations (1):
- Bochner Eye Institute, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No